CLINICAL TRIAL: NCT04843332
Title: Reducing Cancer Disparities Through Innovative Community-Academic Partnership to Advance Access and Delivery of Precision Medicine in Monterey County
Brief Title: Community Health Workers and Precision Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: California Initiative to Advance Precision Medicine (Other); Pacific Cancer Care (Other); The Latino Cancer Institute (Unknown); Cancer Patients Alliance (Unknown)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 59885; OPR18113 (Other Grant/Funding Number: California Initiative to Advance Precision Medicine)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Tumor
Keywords: Precision medicine; Cancer care; lay health worker; community health worker; cancer treatment; patient satisfaction; palliative care; cancer diagnosis; quality of care; tumor testing; End-of-life
MeSH Terms: conditions — Neoplasms; Patient Satisfaction; Death

STUDY DESIGN:
Intervention Model Description: This will be a parallel two-arm randomized controlled trial with the following two arms: (1) usual oncology care or (2) usual oncology care + supplemental community health worker intervention. All participants who consent to the study will be randomized 1:1 into the usual oncology care arm versus the intervention arm. Patients randomized into the intervention arm will be assigned a community health worker who will begin the intervention. Each arm will include 55 participants (total for the study n=110).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Oncology Care (No Intervention): This arm is the control group. They will receive usual oncology care from their regular oncologist and care team with no change in their care plan or treatment as a result of the intervention. Outcomes will be assessed at each of the following times: baseline, 3-months, 6-months, and 12-months.
- Community Health Worker Intervention (Experimental): This arm is the treatment group. Patients randomized into the intervention will be assigned a community health worker who will contact the patient to begin the intervention. They will receive usual oncology care from their regular oncologist and care team but will also receive supplemental support and health education from a community health worker. The lay health worker will assist patients in ensuring that patients discuss the following with their cancer care teams: 1) precision medicine 2) cancer diagnosis and treatment plan 3) adherence to treatments and 3) goals of care and 4) symptom burden. Outcomes will be assessed at each of the following times: baseline, 3-months, 6-months, and 12-months.
  Interventions: Behavioral: Community Health Worker Support

INTERVENTIONS:
Behavioral: Community Health Worker Support — For those in the experimental group, a community health worker will provide health education and support as described in the Community Health Worker Intervention arm.
  Arms: Community Health Worker Intervention

SUMMARY:
The purpose of this randomized controlled trial is to evaluate whether a trained community health worker (CHW) who engages with newly diagnosed patients after a diagnosis of cancer can effectively improve knowledge and receipt of evidence-based precision medicine cancer care services among low-income and minority patients.

DETAILED DESCRIPTION:
The goal of this study is to reduce cancer disparities by improving the knowledge and delivery of evidence-based precision medicine for cancer care. We plan to randomize newly diagnosed patients and those currently under cancer care to either a control arm (usual cancer care alone) versus an intervention arm (layered on top of usual cancer care alone) where patients are assigned to a community health worker who will assist patients in ensuring the following discussions with their care team: 1) precision cancer care 2) cancer diagnosis and treatment plan 2) adherence to treatments and 3) goals of care and symptom burden. A total of 55 participants per study group (total 110) will be recruited in Monterey County from Pacific Cancer Care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with a cancer diagnosis.
* Patients with any relapse or progressive disease (any cancer diagnosis) as identified by imaging or biopsy and confirmed by a physician.
* The patients must be 18 years or older.
* Patients must have the capacity to verbally consent in English or Spanish.
* Patients must be racial/ethnic minorities OR low-income status OR public insurance (Medi-Cal or other) OR have health insurance provided by an agricultural company OR be uninsured

Exclusion Criteria:

* Patients under 18 years of age.
* Inability to consent to the study due to lack of capacity as documented by the referring physician.
* Patients without a newly diagnosed malignancy or patients without relapse of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of precision medicine for cancer care from time of enrollment to 3 months post-enrollment | Time of Enrollment to 3-months post-enrollment
  Using 7 multiple choice items adapted from an 8-item survey tool, Knowledge and Purpose of Molecular Profiling, by Davies et. al., 2020, we will assess knowledge of precision medicine (molecular profiling and tumor testing) for cancer care. All questions are multiple choice. For example one question asks 'tumor testing is helpful for making decisions about future cancer risks,' with answer choices: always, frequently, sometimes, rarely, never, or I don't know. Answers will be scored as number or percent correct.
  Adapted from the following paper: Davies, G., Butow, P., Napier, C. E., Bartley, N., Juraskova, I., Meiser, B., ... & Best, M. C. (2020). Advanced Cancer Patient Knowledge of and Attitudes towards Tumor Molecular Profiling. Translational Oncology, 13(9), 100799.
Knowledge of precision medicine for cancer care | 6-months post-enrollment
  Using 7 multiple choice items adapted from an 8-item survey tool, Knowledge and Purpose of Molecular Profiling, by Davies et. al., 2020, we will assess knowledge of precision medicine (molecular profiling and tumor testing) for cancer care. All questions are multiple choice. For example one question asks 'tumor testing is helpful for making decisions about future cancer risks,' with answer choices: always, frequently, sometimes, rarely, never, or I don't know. Answers will be scored as number or percent correct.
  Adapted from the following paper: Davies, G., Butow, P., Napier, C. E., Bartley, N., Juraskova, I., Meiser, B., ... & Best, M. C. (2020). Advanced Cancer Patient Knowledge of and Attitudes towards Tumor Molecular Profiling. Translational Oncology, 13(9), 100799.
Knowledge of precision medicine for cancer care | 12-months post-enrollment
  Using 7 multiple choice items adapted from an 8-item survey tool, Knowledge and Purpose of Molecular Profiling, by Davies et. al., 2020, we will assess knowledge of precision medicine (molecular profiling and tumor testing) for cancer care. All questions are multiple choice. For example one question asks 'tumor testing is helpful for making decisions about future cancer risks,' with answer choices: always, frequently, sometimes, rarely, never, or I don't know. Answers will be scored as number or percent correct.
  Adapted from the following paper: Davies, G., Butow, P., Napier, C. E., Bartley, N., Juraskova, I., Meiser, B., ... & Best, M. C. (2020). Advanced Cancer Patient Knowledge of and Attitudes towards Tumor Molecular Profiling. Translational Oncology, 13(9), 100799.

SECONDARY OUTCOMES:
Patient activation using the "Patient Activation Measure" survey | 3-months post-enrollment
  Each patient will receive a validated patient activation survey using the "Patient Activation Measure" at enrollment and 3 months after study enrollment. This is a validated measure from Insignia Health. Responses are: disagree strongly, disagree, agree, agree strongly with higher activation correlated with responses of agree and agree strongly. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-10, minimum score is 0 (if all not-applicable) and maximum is 40. Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining "Behaviors and Pushing Further. Scores for each group will be averaged at 3 months after study enrollment.
Patient activation using the "Patient Activation Measure" survey | 6-months post-enrollment
  Each patient will receive a validated patient activation survey using the "Patient Activation Measure" at enrollment and 6 months after study enrollment. This is a validated measure from Insignia Health. Responses are: disagree strongly, disagree, agree, agree strongly with higher activation correlated with responses of agree and agree strongly. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-10, minimum score is 0 (if all not-applicable) and maximum is 40. Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining "Behaviors and Pushing Further. Scores for each group will be averaged at 6 months after study enrollment.
Patient activation using the "Patient Activation Measure" survey | 12-months post-enrollment
  Each patient will receive a validated patient activation survey using the "Patient Activation Measure" at enrollment and 12 months after study enrollment. This is a validated measure from Insignia Health. Responses are: disagree strongly, disagree, agree, agree strongly with higher activation correlated with responses of agree and agree strongly. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-10, minimum score is 0 (if all not-applicable) and maximum is 40. Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining "Behaviors and Pushing Further. Scores for each group will be averaged at 12 months after study enrollment.
Patient Satisfaction With Decision measured with the "Satisfaction with Decision Instrument" | 3-months post-enrollment
  Each patient will receive an adapted version of the 6-item Satisfaction with Decision Instrument at 3 months after study enrollment. Responses are "completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, or completely agree," with 1=completely disagree and 6= completely agree. Higher scores indicate greater levels of satisfaction. Minimum score is 9, maximum is 54. Responses for each group will be assessed at 3 months after study enrollment. The measure is adapted from: Holmes-Rovner, M., Kroll, J., Schmitt, N., Rovner, D. R., Breer, M. L., Rothert, M. L., ... & Talarczyk, G. (1996). Patient satisfaction with health care decisions: the satisfaction with decision scale. Medical Decision Making, 16(1), 58-64.
Patient Satisfaction With Decision measured with the "Satisfaction with Decision Instrument" | 6-months post-enrollment
  Each patient will receive an adapted version of the 6-item Satisfaction with Decision Instrument at 6 months after study enrollment. Responses are "completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, or completely agree," with 1=completely disagree and 6= completely agree. Higher scores indicate greater levels of satisfaction. Minimum score is 9, maximum is 54. Responses for each group will be assessed at 3 months after study enrollment. The measure is adapted from: Holmes-Rovner, M., Kroll, J., Schmitt, N., Rovner, D. R., Breer, M. L., Rothert, M. L., ... & Talarczyk, G. (1996). Patient satisfaction with health care decisions: the satisfaction with decision scale. Medical Decision Making, 16(1), 58-64.
7. Patient Satisfaction With Decision measured with the "Satisfaction with Decision Instrument" | 12-months post-enrollment
  Each patient will receive an adapted version of the 6-item Satisfaction with Decision Instrument at 12 months after study enrollment. Responses are "completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, or completely agree," with 1=completely disagree and 6= completely agree. Higher scores indicate greater levels of satisfaction. Minimum score is 9, maximum is 54. Responses for each group will be assessed at 3 months after study enrollment. The measure is adapted from: Holmes-Rovner, M., Kroll, J., Schmitt, N., Rovner, D. R., Breer, M. L., Rothert, M. L., ... & Talarczyk, G. (1996). Patient satisfaction with health care decisions: the satisfaction with decision scale. Medical Decision Making, 16(1), 58-64.
Palliative Care Utilization (Chart Review) | 12 months post-enrollment
  Medical record review for quantity of use of any palliative care, any hospice, any chemotherapy, any radiotherapy, or any surgery.
Patient Quality of Life Using the "Functional Assessment of Cancer Therapy - General Survey" | Time of enrollment to 3-months post-enrollment
  Each patient will the validated "Functional Assessment of Cancer Therapy - General Survey (FACT-G), " which is a 27-item survey with response options including: not at all, a little bit, somewhat, quite a bit, or very much. Five items also allow for a response of 'prefer not to answer.' Scoring for the FACT-G will be done in accordance with the FACT-G Scoring Guidelines (Version 4), available here: https://www.facit.org/measures-scoring-downloads/fact-g-scoring-downloads . In summary, scoring is for four subscales included within the survey, including (1) Physical Well-Being (score range: 0-28), (2) Social Family Well-Being (score range: 0-28), (3) Emotional Well-Being (score range: 0-24), and (4) Functional Well-Being (score range: 0-28). A total score is created from the sum of the subscale scores and has a minimum of zero and maximum of 108, where a higher score indicates greater quality of life. We will measure the change in quality of life at baseline to 3 months.
Patient Quality of Life Using the "Functional Assessment of Cancer Therapy - General Survey" | 6 months post-enrollment
  Each patient will the validated "Functional Assessment of Cancer Therapy - General Survey (FACT-G), " which is a 27-item survey with response options including: not at all, a little bit, somewhat, quite a bit, or very much. Five items also allow for a response of 'prefer not to answer.' Scoring for the FACT-G will be done in accordance with the FACT-G Scoring Guidelines (Version 4), available here: https://www.facit.org/measures-scoring-downloads/fact-g-scoring-downloads . In summary, scoring is for four subscales included within the survey, including (1) Physical Well-Being (score range: 0-28), (2) Social Family Well-Being (score range: 0-28), (3) Emotional Well-Being (score range: 0-24), and (4) Functional Well-Being (score range: 0-28). A total score is created from the sum of the subscale scores and has a minimum of zero and maximum of 108, where a higher score indicates greater quality of life. We will measure the change in quality of life at baseline to 6 months.
Patient Quality of Life Using the "Functional Assessment of Cancer Therapy - General Survey" | 12 months post-enrollment
  Each patient will the validated "Functional Assessment of Cancer Therapy - General Survey (FACT-G), " which is a 27-item survey with response options including: not at all, a little bit, somewhat, quite a bit, or very much. Five items also allow for a response of 'prefer not to answer.' Scoring for the FACT-G will be done in accordance with the FACT-G Scoring Guidelines (Version 4), available here: https://www.facit.org/measures-scoring-downloads/fact-g-scoring-downloads . In summary, scoring is for four subscales included within the survey, including (1) Physical Well-Being (score range: 0-28), (2) Social Family Well-Being (score range: 0-28), (3) Emotional Well-Being (score range: 0-24), and (4) Functional Well-Being (score range: 0-28). A total score is created from the sum of the subscale scores and has a minimum of zero and maximum of 108, where a higher score indicates greater quality of life. We will measure the change in quality of life at baseline to 12 months.
Prognosis & Treatment Preference | 6 months post-enrollment
  Patients will answer 4 multiple choice items to assess understanding of their prognosis and their treatment preferences. These items are not part of a named tool. They are adapted from the prognosis and treatment preference items developed by Weeks et al. (1998).
  1. Is your cancer curable? Response options (ROs): Yes, No, I don't know
  2. How long do most patients with your disease live on average? ROs: Less than 6 months, 6 months - 2 years, More than 2 years, I don't know
  3. The goal of my cancer treatment is to: (select all that apply) ROs: Cure my disease, help me feel better, extend my life, I don't know
  4. Would you prefer a course of treatment that focuses on extending life as much as possible, even if it means having more pain and discomfort, or would you want a plan of care that focuses on relieving pain and discomfort, even if that means not living as long? ROs: Extend life as much as possible, relieve pain or discomfort as much as possible, I don't know
Prognosis & Treatment Preference | 12 months post-enrollment
  Patients will answer 4 multiple choice items to assess understanding of their prognosis and their treatment preferences. These items are not part of a named tool. They are adapted from the prognosis and treatment preference items developed by Weeks et al. (1998).
  1. Is your cancer curable? Response options (ROs): Yes, No, I don't know
  2. How long do most patients with your disease live on average? ROs: Less than 6 months, 6 months - 2 years, More than 2 years, I don't know
  3. The goal of my cancer treatment is to: (select all that apply) ROs: Cure my disease, help me feel better, extend my life, I don't know
  4. Would you prefer a course of treatment that focuses on extending life as much as possible, even if it means having more pain and discomfort, or would you want a plan of care that focuses on relieving pain and discomfort, even if that means not living as long? ROs: Extend life as much as possible, relieve pain or discomfort as much as possible, I don't know
Prognosis & Treatment Preference | 3 months post-enrollment
  Patients will answer 4 multiple choice items to assess understanding of their prognosis and their treatment preferences. These items are not part of a named tool. They are adapted from the prognosis and treatment preference items developed by Weeks et al. (1998).
  1. Is your cancer curable? Response options (ROs): Yes, No, I don't know
  2. How long do most patients with your disease live on average? ROs: Less than 6 months, 6 months - 2 years, More than 2 years, I don't know
  3. The goal of my cancer treatment is to: (select all that apply) ROs: Cure my disease, help me feel better, extend my life, I don't know
  4. Would you prefer a course of treatment that focuses on extending life as much as possible, even if it means having more pain and discomfort, or would you want a plan of care that focuses on relieving pain and discomfort, even if that means not living as long? ROs: Extend life as much as possible, relieve pain or discomfort as much as possible, I don't know
Receipt of Molecular Profile and Genomic Testing | 12 months post-enrollment
  We will look at the percent of patients with receipt of molecular tumor profile and genomic testing (evidence-based treatment)
Emergency Department Visit (Chart Review) | 12 months post-enrollment
  Emergency Department Use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Hospitalization Visit (Chart Review) | 12 months post-enrollment
  Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Study data will not be shared with researchers outside of this project.

REFERENCES:
- [Background] Davies G, Butow P, Napier CE, Bartley N, Juraskova I, Meiser B, Ballinger ML, Thomas DM, Schlub TE, Best MC; members of the PiGeOn Project. Advanced Cancer Patient Knowledge of and Attitudes towards Tumor Molecular Profiling. Transl Oncol. 2020 Sep;13(9):100799. doi: 10.1016/j.tranon.2020.100799. Epub 2020 May 22. PMID 32450551
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] Weeks JC, Cook EF, O'Day SJ, Peterson LM, Wenger N, Reding D, Harrell FE, Kussin P, Dawson NV, Connors AF Jr, Lynn J, Phillips RS. Relationship between cancer patients' predictions of prognosis and their treatment preferences. JAMA. 1998 Jun 3;279(21):1709-14. doi: 10.1001/jama.279.21.1709. PMID 9624023
- [Derived] Rodriguez GM, Wood EH, Xiao L, Duron Y, O'Brien D, Koontz Z, Rosas LG, Patel MI. Community health workers and precision medicine: A randomized controlled trial. Contemp Clin Trials. 2022 Oct;121:106906. doi: 10.1016/j.cct.2022.106906. Epub 2022 Sep 6. PMID 36084898
- See also: Scoring Guide for FACT-G — https://www.facit.org/measures-scoring-downloads/fact-g-scoring-downloads